CLINICAL TRIAL: NCT03926858
Title: Patient-reported Outcomes of Postsurgical Pain and Health Related Quality of Life, a Multi-centered, Prospective, Observational, Cohort Study
Brief Title: Patient-reported Outcomes of Postsurgical Pain and Health Related Quality of Life
Acronym: HRQoL
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Director of department of anesthesiology and pain management, Peking University People's Hospital
Other Study IDs: 2018PHB229-01
Record Dates: First submitted 2019-04-17; First posted 2019-04-25 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Post Surgical Pain
Keywords: post-surgical pain; health-related quality of life
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will investigate the impact of post-surgical pain (PSP) on health related quality of life (HRQoL) within the first six months following surgery using patient-reported outcome (PRO) measures, and to investigate medical recovery measures such as ambulation and oral feeding time as secondary outcomes.

DETAILED DESCRIPTION:
Pain and recovery after surgery are extremely concerned by patients undergoing surgery. Though it is important to understand the recovery course of postsurgical pain and recovery, most previous studies just focused on one specific time point, and the results were inconsistent.

To investigate the impact of PSP on HRQoL within the first six months following surgery using PRO measures, patients undergoing several specific surgeries will be interviewed. Patients' medical charts will be reviewed by investigators to record sociodemographic and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing general or regional anesthesia
* Hospitalized for at least 24 hours after surgery

Exclusion Criteria:

* Existing diagnoses of psychiatric pathology
* Surgery cancellation
* Unable to give informed consent
* Unable to read and write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing the following procedures: breast surgery, thoracic surgery, abdominal surgery, orthopedic surgery.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Health related quality of life(HRQoL) | up to 6 months after surgery
  HRQoL is measured with EuroQol five-dimensional questionnaire(EQ-5D).
Pain after surgery | up to 6 months after surgery
  Postsurgical pain is measured with the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) .

SECONDARY OUTCOMES:
ambulation time | up to 30 days after surgery
  the first time when patients can get off of bed and walk after surgery
oral feeding time | up to 30 days after surgery
  the first time when patients begin oral feeding after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, PhD, Principal Investigator — Peking University People's Hospital; Xiumei Gao, MD, Study Director — Xiyuan Hospital; Jingzhi Liu, Study Director — Tianjin Medical University Second Hospital; Guanghe Si, MD, Study Director — Songyuan Central Hospital; Yaying Xie, Study Director — The Affiliated Hospital of Inner Mongolia Medical University; Jun Yan, Study Director — Huhhot First Hospital; Aizhi Li, Study Director — Yantai Yuhuangding Hospital; Weiwei Zhang, MD, Study Director — Shanxi Provincial People's Hospital; Zhenhua Qu, MD, Study Director — Xingtai People's Hospital; Ying Wang, MD, Study Director — The First Affiliated Hospital of Zhengzhou University; Hongguang Bao, Study Director — The First Affiliated Hospital with Nanjing Medical University; Weidong Gu, Study Director — Huadong Hospital; Fan Tao, Study Director — Red Cross Hospital, Hangzhou, China; Hongwei Wang, Study Director — Zhejiang Provincial Tongde Hospital; Xianwei Zhang, Study Director — Tongji Hospital; Qingpeng Dong, Study Director — The Third People's Hospital of Hubei Province; Qin Liao, Study Director — The Third Xiangya Hospital of Central South University; Caiping Liao, Study Director — The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine; Haihua Shu, Study Director — Guangdong Second Provincial Central Hospital; Zhijun Chen, Study Director — Guilin Medical University, China; Yubo Xie, Study Director — First Affiliated Hospital of Guangxi Medical University; Bangxiang Yang, Study Director — West China Hospital; Hui Huang, Study Director — The Ninth People's Hospital of Chongqing; Xiang Shen, Study Director — The First People's Hospital of Liangshan Yi Autonomous Prefecture; Shaoxing Dong, Study Director — People's Hospital of Yuxi; Yimei Li, Study Director — First Affiliated Hospital of Xinjiang Medical University
Locations (23):
- China (23):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Third People's Hospital of Hubei Province, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - The First Hospital of Changsha, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Baotou, Inner Mongolia
  - Huhhot First Hospital, Hohhot, Inner Mongolia
  - Nanjing First Hospital, Nanyang, Jiangsu
  - Songyuan Central Hospital, Songyuan, Jilin
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First People's Hospital of Liangshan Yi Autonomous Prefecture, Liangshan, Yunan
  - People's Hospital of Yuxi, Yuxi, Yunnan
  - Hangzhou Red Cross Hospital, Hangzhou, Zhejiang
  - Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Xiyuan Hospital, Beijing
  - The Ninth People's Hospital of Chongqing, Chongqing
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - The Second Hospital of Tianjin Medical University, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Taylor RS, Ullrich K, Regan S, Broussard C, Schwenkglenks M, Taylor RJ, Gordon DB, Zaslansky R, Meissner W, Rothaug J, Langford R; PAIN-OUT investigators. The impact of early postoperative pain on health-related quality of life. Pain Pract. 2013 Sep;13(7):515-23. doi: 10.1111/papr.12026. Epub 2012 Dec 23. PMID 23279591
- [Derived] Zhang Q, Wu Y, Hong S, Feng Y. Trajectory of worst pain within the first two weeks following pelvic and sacral tumor surgery and long-term outcome: a pilot observational prospective cohort study. BMC Anesthesiol. 2023 Mar 9;23(1):73. doi: 10.1186/s12871-023-02033-z. PMID 36894887